CLINICAL TRIAL: NCT02054091
Title: Bovine Colostrum as Nutrition for Preterm Infants in the First Days of Life: A Pilot Feasibility Study
Brief Title: Feeding Bovine Colostrum to Preterm Infants
Acronym: PreColos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Per Torp Sangild (Other)
Responsible Party: Sponsor-Investigator, Per Torp Sangild, Professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H-3-2013-136
Record Dates: First submitted 2014-01-21; First posted 2014-02-04 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Feeding Intolerance; Extrauterine Growth Retardation; Necrotizing Enterocolitis; Sepsis; Meningitis
Keywords: Preterm infants; Bovine colostrum; Feeding intolerance; Postnatal growth; Intestinal maturation; Necrotizing enterocolitis
MeSH Terms: conditions — Enterocolitis, Necrotizing; Sepsis; Meningitis

STUDY DESIGN:
Intervention Model Description: Single group for first 12 infants RCT for next 40 infants
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): Infants are fed according to the standard feeding practices at each hospital. At FWCH & SBMCH babies are fed infant formula supplemented to mother's own milk (if avaible), and at RH, babies are fed donor milk supplemented to Mother'w own milk (if avaible).
- Colostrum group (Experimental): Infants are fed bovine colostrum supplemented to mother's own milk (if avaible) for max. 10 days at RH and 14 days at FWCH & SBMCH.
  Interventions: Dietary Supplement: Bovine colostrum

INTERVENTIONS:
Dietary Supplement: Bovine colostrum — The BC powder to be used in this study is donated from a Danish company, Biofiber Damino. The raw colostrum used for production is collected within 1-2 milking from healthy Danish dairy cows (Danish Holstein). Antibiotic residues are screened upon collection and those tested positive are not used for production. Intact colostrum is pasteurized, low temperature spray-dried, and sterilized by γ-irradiation.
  Other Names: Cow's colostrum
  Arms: Colostrum group

SUMMARY:
Feeding preterm infants is of great challenge in the NICUs. Mother's own milk is considered as the best for the digestive system followed by donor milk. Preterm infant formula is related to more feeding problems and other gut complications in these babies, such as necrotizing enterocolitis. Bovine colostrum contains higher amounts of protein, growth factors and immuno-regulatory components (e.g. immunoglobulins), which has been used in many other situations to promote health. The investigators plan to give bovine colostrum to preterm infants with birth weights between 1000 and 1800 g, or born between 27+0 and 32+6 weeks of gestational age, in order to promote feeding and intestinal health in these babies. This current study is a feasibility pilot study and the investigators hypothesized that supplementing BC to MM (if available) is safe and tolerable when used within the first 10-14 days of life in preterm infants.

DETAILED DESCRIPTION:
Preterm birth (<37 weeks gestation) occurs in 10% of all pregnancies worldwide and the optimal way to feed a newborn preterm infant, when breast-feeding is impossible, is not clear. Excessive enteral feeding predisposes to various complications and necrotizing enterocolitis (NEC) that occur in 7% of preterm infants born with less than 1500 g body weight. Early feeding with small volumes of milk is applied to promote GIT maturation and add some nutrients and energy. It is assumed that early feeding allows more rapid advancement to full enteral feeding (EN, e.g 120-160 ml/kg/d) and weaning from parenteral nutrition (PN). This is important to reduce PN-related complications (e.g. sepsis) and to better stimulate body and organ (e.g. gut, brain) development. However, it remains unclear what is the best milk diet when mother's own milk (MM) is not available. Infant formula (IF) and banked human donor milk (DM) are the most frequently used alternatives to MM. MM is superior to IF in promoting feeding tolerance, intestinal function, and NEC resistance in preterm infants. Feeding with DM is also believed to be beneficial, relative to IF, although this pasteurized milk obtained from mothers later in lactation may be less beneficial, relative to the first milk, colostrum. There are differences in the amount and composition between human colostrum and bovine colostrum (BC), but relative to mature human milk, BC contains higher amounts of protein, growth factors and immuno-regulatory components (e.g. immunoglobulins). Large amount of protein in BC provides higher enteral protein intake and may enable a reduction in the use of PN and central venous catheters, and hereby reduced risk of infection. Also this may lead to reduced weight loss and improved growth of the brain and the body. In addition, maturational and NEC-protective effects of BC have repeatedly been documented in preterm pigs when BC is used as the first diet after birth. The investigators therefore plan to investigate whether using BC as nutrition for preterm infants in the first weeks of life is safe, tolerable, and helps to provide nutrients and gut maturation , when MM is not in sufficient amounts or not available.

ELIGIBILITY:
Inclusion Criteria:

* FWCH & SBMCH: Preterm infants with birth weights between 1000 and 1800 g, delivered at FWCH & SBMCH, or transferred from other hospitals within 24 h of birth and without any enteral feeding.

RH & HH: Preterm infants less than 24 hours of age, between 27+0 and 32+6 weeks of gestation, delivered at RH &HH , or transferred from other hospitals within the first 24 h after birth.

* Signed parental consent

Exclusion Criteria:

* Major congenital anomalies or birth defects
* Congenital infection
* Perinatal asphyxia
* Gestational age at birth < 28 weeks (FWCH & SBMCH)
* Extremely SGA infant (weight SD score < -3 SD)
* Need for mechanical ventilation or cardiovascular support before first BC feeding

Max Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the tolerability of bovine colostrum feeding | From birth until the recruited subject reaches postmenstrual age at 37 weeks or discharge home, whichever comes first
  The main purpose of this feasibility pilot study is to investigate whether preterm infants can tolerate bovine colostrum as their first nutrition supplemented to mother's own milk (if available). Presence of feeding intolerance is defined as at any time when feeding is withheld by the neonatologists from day 1-7 and from day 8-14.

SECONDARY OUTCOMES:
Anthropometry data | Weekly measured from birth until the recruited subject reaches postmenstrual age at 37 weeks or discharge home, whichever comes first
  Body weight, body length, and head circumference are measured as anthropometry data
Days to regain birth weight | From birth until the recruited subject reaches postmenstrual age at 37 weeks or discharge home, whichever comes first
Days on parenteral nutrition | From birth until the recruited subject reaches postmenstrual age at 37 weeks or discharge home, whichever comes first
  Days on PN are the total number of days that a participant receiving any i.v. nutrients other than glucose.
Time to full enteral feeding | From birth until the recruited subject reaches postmenstrual age at 37 weeks or discharge home, whichever comes first
  Full enteral feeding is defined as participants receiving 160ml/kg/d at copenhagen site, or more than 120 ml/kg/d at Chinese sites for a consecutive period of 72 hours.
Combined incidence of serious infections and NEC | From birth until the recruited subject reaches postmenstrual age at 37 weeks or discharge home, whichever comes first
  Serious infections/NEC includes sepsis and meningitis, according the diagnostic criteria at each hospital, and Bell stage II or III NEC.
Plasma citrulline level | On day 7±1 at RH & HH and on day 7±1 and 14±1 at FWCH & SBMCH
  Citrulline concentration is measured in plasma as a biomarker for absorptive enterocyte mass and/or function
Lactase activity and intestinal permeability | On day 7±1
  Lactase activity and intestinal permeability is measured non-invasively by measuring the urinary ratio of lactulose/lactose, and lactulose/mannitol after the three sugars are administered.

OTHER OUTCOMES:
Routine blood tests | On day 7±1 at RH & HH and on day 7±1 and 14±1 at FWCH & SBMCH
  Routine blood tests include blood gas analysis, liver enzymes, BUN, creatinine, Na, K, and phosphate.
Plasma amino acid composition | On day 7±1 at RH & HH and on day 7±1 and 14±1 at FWCH & SBMCH
  Plasma amino acids will be analyzed at each hospital to investigate whether BC feeding provides a normal range of plasma amino acid pattern.
Plasma bovine IgG level | On day 7±1 at RH for phase A and B
  The concentration of intact bovine IgG will be measured in the plasma samples from the participants who receive BC supplementation, in order to investigate how much intact bovine IgG is absorbed from the intestine and circulating in the blood. This will only be measured in the participants at RH due to practical reasons.
Fecal bovine IgG | On day 7±1 at RH & HH and day 7±1 and 14±1 days
  The concentration of intact bovine IgG will be measured in the fecal samples from participants who receive BC supplementation, in order to investigate whether bovine IgG can survive digestion.
Fecal short chain fatty acids (SCFAs) | On day 7±1 at RH & HH and day 7±1 and 14±1 days
  Fecal SCFAs will be measured as an indicator of bacterial fermentation of the unabsorbed nutrients in the colon.
Fecal microbiota composition | On day 7±1 at RH & HH and day 7±1 and 14±1 days
  Microbiota composition in fecal samples will be determined using non-culture-based techniques

CONTACTS AND LOCATIONS:
Overall Officials: Per T. Sangild, PhD, Study Director — +45 35 33 26 98
Locations (4):
- China (2):
  - Foshan Women and Children's Hospital (FWCH), Foshan, Guangdong
  - Shenzheng Baoan Maternity and Child Healthcare Hospital (SBMCH), Shenzhen, Guangdong
- Denmark (2):
  - Rigshospitalet (RH), Copenhagen
  - Hvidovre Hospital (HH), Hvidovre

REFERENCES:
- See also: The current clinical trial is a part of the NEOMUNE project. — http://neomune.ku.dk/